CLINICAL TRIAL: NCT00303875
Title: RENEW: Reach Out to Enhance Wellness in Older Survivors
Brief Title: Exercise and Dietary Counseling in Improving Physical Activity, Nutrition, and Quality of Life in Older Long-Term Cancer Survivors Who Are Overweight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00012963; DUMC-5477-03-12R0ER; DUMC-5477-04-12R1ER; CDR0000460231 (Other: NCI)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2013-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait-list control (No Intervention): Wait-list control received diet & exercise counseling during year 2 as a courtesy
- Lifestyle counseling (Experimental): subjects randomized to receive diet & exercise counseling for one year
  Interventions: Behavioral: behavioral dietary and exercise intervention

INTERVENTIONS:
Behavioral: behavioral dietary and exercise intervention
  Arms: Lifestyle counseling

SUMMARY:
RATIONALE: Exercise and dietary counseling may improve physical activity, nutrition, and quality of life in older long-term cancer survivors who are overweight.

PURPOSE: This randomized clinical trial is studying two different schedules of exercise and dietary counseling to compare how well they work in improving physical activity, nutrition, and quality of life in older long-term cancer survivors who are overweight.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the physical function over 1 year of overweight older long-term cancer survivors assigned to immediate vs delayed exercise and dietary counseling.

Secondary

* Compare physical activity, saturated fat and vegetable and fruit intake, body mass index, depression, and general health and well being of experimental arm patients vs control arm patients.
* Evaluate self-efficacy, social support, comorbidity, cancer-type, and gender as factors associated with program efficacy.
* Determine the functional decline over a 2-year period in patients who undergo immediate vs delayed intervention.
* Characterize the mathematical form, over a 2-year period, of physical functioning trajectories among older cancer survivors, including determining if the intervention effects are durable in those who receive the intervention initially and whether "catch-up" is possible in the delayed intervention arm.

OUTLINE: This is a randomized study. Patients are stratified according to cancer type (colorectal vs breast or prostate), sex, age (65-74 years vs 75 years and over), and race (white vs non-white). Patients are randomized to 1 of 2 intervention arms.

* Arm I (immediate intervention): Patients receive a personalized notebook of diet and exercise information, exercise equipment, and logbooks to record food intake and exercise behaviors. Patients undergo 20-minute telephone discussions with a health counselor once weekly for 3 weeks, every 2 weeks for 2 months, and then monthly for up to 1 year for a total of 15 sessions. Patients also undergo a 5-minute telephone survey to assess health every 3 months.
* Arm II (delayed intervention): Patients undergo intervention as in arm I after a 1-year waiting period.

After completion of study intervention, patients are followed periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 640 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed colorectal, prostate, or female breast cancer

  * At least 5 years beyond date of diagnosis with no clinical evidence of progressive disease or second primaries
* Body mass index ≥ 25 kg/m^2 and < 40 kg/m^2
* Currently exercising < 150 minutes/week
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No serious intercurrent medical condition or disability that could preclude study treatment, including any of the following:

  * Severe orthopedic condition or scheduled hip or knee replacement within the next 6 months
  * Paralysis
  * End-stage renal disease
  * Dementia
  * Unstable angina
  * Heart attack, congestive heart failure, or pulmonary condition that required oxygen or hospitalization within the past 6 months
* Ability to read, write, and speak English

PRIOR CONCURRENT THERAPY:

* No concurrent warfarin

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 641 (Actual)
Dates: Start 2003-12; Primary Completion 2008-06 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Physical function as assessed by Short-Form Health Survey (SF-36) with physical function subscale and late effects lower body subscales at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.

SECONDARY OUTCOMES:
Quality of life as assessed by SF-36 at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Physical activity as assessed by Community Healthy Activities Model Program for Seniors (CHAMPS) at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Dietary intake as assessed by 2-day dietary recalls at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Body weight status as assessed by body mass index at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Depression and/or anxiety as assessed by Hospital Anxiety Depression Scale at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Self-efficacy for exercise and dietary change assessed by self-efficacy algorithms at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.
Stage of readiness for exercise and dietary change as assessed by the stage of change algorithms at baseline and years 1 and 2 following study completion | one year
  one year for intervention subjects - in year two, wait listed controls received intervention and the intervention subjects were followed.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Result] Demark-Wahnefried W, Morey MC, Sloane R, Snyder DC, Miller PE, Hartman TJ, Cohen HJ. Reach out to enhance wellness home-based diet-exercise intervention promotes reproducible and sustainable long-term improvements in health behaviors, body weight, and physical functioning in older, overweight/obese cancer survivors. J Clin Oncol. 2012 Jul 1;30(19):2354-61. doi: 10.1200/JCO.2011.40.0895. Epub 2012 May 21. PMID 22614994
- [Result] Miller PE, Morey MC, Hartman TJ, Snyder DC, Sloane R, Cohen HJ, Demark-Wahnefried W. Dietary patterns differ between urban and rural older, long-term survivors of breast, prostate, and colorectal cancer and are associated with body mass index. J Acad Nutr Diet. 2012 Jun;112(6):824-31, 831.e1. doi: 10.1016/j.jand.2012.02.021. PMID 22709810
- [Result] Mosher CE, Sloane R, Morey MC, Snyder DC, Cohen HJ, Miller PE, Demark-Wahnefried W. Associations between lifestyle factors and quality of life among older long-term breast, prostate, and colorectal cancer survivors. Cancer. 2009 Sep 1;115(17):4001-9. doi: 10.1002/cncr.24436. PMID 19637244
- [Result] Morey MC, Snyder DC, Sloane R, Cohen HJ, Peterson B, Hartman TJ, Miller P, Mitchell DC, Demark-Wahnefried W. Effects of home-based diet and exercise on functional outcomes among older, overweight long-term cancer survivors: RENEW: a randomized controlled trial. JAMA. 2009 May 13;301(18):1883-91. doi: 10.1001/jama.2009.643. PMID 19436015
- [Result] Snyder DC, Morey MC, Sloane R, Stull V, Cohen HJ, Peterson B, Pieper C, Hartman TJ, Miller PE, Mitchell DC, Demark-Wahnefried W. Reach out to ENhancE Wellness in Older Cancer Survivors (RENEW): design, methods and recruitment challenges of a home-based exercise and diet intervention to improve physical function among long-term survivors of breast, prostate, and colorectal cancer. Psychooncology. 2009 Apr;18(4):429-39. doi: 10.1002/pon.1491. PMID 19117329
- [Result] Morey MC, Blair CK, Sloane R, Cohen HJ, Snyder DC, Demark-Wahnefried W. Group trajectory analysis helps to identify older cancer survivors who benefit from distance-based lifestyle interventions. Cancer. 2015 Dec 15;121(24):4433-40. doi: 10.1002/cncr.29684. Epub 2015 Oct 29. PMID 26512712
- [Result] Winger JG, Mosher CE, Rand KL, Morey MC, Snyder DC, Demark-Wahnefried W. Diet and exercise intervention adherence and health-related outcomes among older long-term breast, prostate, and colorectal cancer survivors. Ann Behav Med. 2014 Oct;48(2):235-45. doi: 10.1007/s12160-014-9598-7. PMID 24648018
- [Result] Blair CK, Morey MC, Desmond RA, Cohen HJ, Sloane R, Snyder DC, Demark-Wahnefried W. Light-intensity activity attenuates functional decline in older cancer survivors. Med Sci Sports Exerc. 2014 Jul;46(7):1375-83. doi: 10.1249/MSS.0000000000000241. PMID 24389524
- [Result] Demark-Wahnefried W, Morey MC, Sloane R, Snyder DC, Cohen HJ. Promoting healthy lifestyles in older cancer survivors to improve health and preserve function. J Am Geriatr Soc. 2009 Nov;57 Suppl 2(Suppl 2):S262-4. doi: 10.1111/j.1532-5415.2009.02507.x. PMID 20122025
- [Result] Miller P, Demark-Wahnefried W, Snyder DC, Sloane R, Morey MC, Cohen H, Kranz S, Mitchell DC, Hartman TJ. Dietary supplement use among elderly, long-term cancer survivors. J Cancer Surviv. 2008 Sep;2(3):138-48. doi: 10.1007/s11764-008-0060-3. Epub 2008 Jul 11. PMID 18792788